CLINICAL TRIAL: NCT04706858
Title: Integrative Personal Omics Profiling for Dynamic Molecular Phenotypes Monitoring During Fiber Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Snyder, Chair, Dept. of Genetics, Stanford University
Allocation: Not Applicable | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: 1636
Record Dates: First submitted 2020-12-03; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Prebiotics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to start fiber supplementation with one type of fiber for three weeks. After a washout period, they will supplement with the second type of fiber for an additional 3 weeks.The third cycle will be the same for all participants and they will supplement with a mix of 5 fibers for 3 weeks.
Who Masked: Participant
Masking Description: Participant will be given the unlabeled fiber supplement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Dietary fiber supplementation — Randomization to the order of first fiber: either inulin or arabinoxylan. Third cycle will include a mix of 5 fibers: inulin, arabinoxylan, resistant starch, glucomannan, and acacia gum.

SUMMARY:
The investigators propose a comprehensive, multiomic study that will integrate longitudinal data associating changes in specific gut bacteria and host in response to prebiotic fiber supplementation. These data will guide the development of an integrative biological signature relating bacterial-derived metabolites with biological outcome in the host.

DETAILED DESCRIPTION:
With this study, the investigators propose to assemble a cohort of healthy individuals that will receive prebiotic supplementation, during comprehensive, longitudinal characterization of the microbiota and host changes with clinical markers and multiple omics assays. These multiomic data will then be integrated, generating unique biological signatures that define the role that microbial metabolites from specific bacteria play in host biological activity. Through this study the investigators expect to gain a detailed and clear understanding of the physiological changes, at the mechanistic level, that occur in the microbiome and host in response to dietary supplementation with prebiotic fiber.

ELIGIBILITY:
Inclusion Criteria:

* Good general health

Exclusion Criteria:

* Fasting Blood Sugar >126 mg/dL
* Triglycerides >400 mg/dL
* Uncontrolled hypertension
* Vascular disease
* Chronic inflammatory conditions
* Major organ disease
* Heavy alcohol use
* Pregnancy/lactation
* Prior bariatric surgery
* Active psychiatric disease
* Use of medication known to affect carbohydrate or lipid metabolism
* Active eating disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Lipid profile changes in response to prebiotic intervention | 3 years
  Analysis of changes in the the lipid profile of participants on the prebiotic intervention. Measured lipids in mg/dL include total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides.
Mapping of microbiota changes in response to prebiotic intervention | 3 years
  A detailed map of microbes and microbial gene expression changes during the intervention will be developed.
  Microbiota complexity in fecal samples will be determined by shotgun metagenomic sequencing. Novel microbes and gene pathways will be identified by de novo assemble of whole fecal metagenomes.

SECONDARY OUTCOMES:
Comprehensive metagenome profile during prebiotic intervention | 3 years
  Changes in host (human) metagenome profile during the prebiotic intervention will be determined. Stool DNA Sequences are analyzed using the Humann2 and Metaphlan pipelines to generate pathway coverage values, gene families abundances, and taxa abundances {Franzosa, 2018}. These are mapped to the Human Microbiome Project database for alignment.
Comprehensive transcriptome profile during prebiotic intervention | 3 years
  Changes in host (human) transcriptome profile during the prebiotic intervention will be determined. RNA isolated from PBMC samples reads are aligned to hg38 using the program Spliced Transcripts Alignment to a Reference (STAR). Transcript abundance is calculated using RNA-Seq by Expectation Maximization (RSEM). Normalization of transcript frequency and pairwise statistics measuring differences in transcript frequency between time points are calculated using the software package for R from Bioconductor (DESeq2).
Comprehensive metabolome profile during prebiotic intervention | 3 years
  Changes in host (human) metabolome profile during the prebiotic intervention will be determined. Plasma metabolites are run in mass spectrometers columns (HILIC and RPLC separation in both positive and negative ionization modes). MetID and our MS/MS data are used to identify 12740 metabolites with confidence levels ranging from 1-3, where 1 matches MS/MS, retention time and m/z from standards on our platform, 2 has MS/MS and m/z matches from a database, and 3 matches the m/z of a database.
Comprehensive cytokine profile during prebiotic intervention | 3 years
  Changes in host (human) cytokine profile during the prebiotic intervention will be determined. Cytokines are profiled using a Luminex xMAP cytokine profiling system at the Stanford Human Immune Monitoring Center. This involves attaching antibodies specific to cytokines to beads using a capture molecule. The fluorescent molecules are attached to the cytokines, and fluorescence is used as the measure of cytokine abundance.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No